CLINICAL TRIAL: NCT01352546
Title: Open Label, Single Center, Pilot Study of the Use of BOTOX Injections, Sensorcaine Injections and Progressive Dilation Under Anesthesia for the Treatment of Primary Vaginismus
Brief Title: Botox Injection for Treatment of Vaginismus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Plastic Surgery Professional Association (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Peter T. Pacik, MD, FACS, Medical director Plastic Surgery Professional Association, Plastic Surgery Professional Association
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTX-PV-01
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Vaginismus
Keywords: vaginismus; painful sex; painful intercourse; dyspareunia; inability to have intercourse; inability to consummate marriage; vaginal spasm; "hitting a wall"; pain during sex; pain during intercourse; burning with intercourse
MeSH Terms: conditions — Vaginismus; Dyspareunia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BOTOX (Experimental): intravaginal Botox injections and progressive dilation under anesthesia to cure vaginismus.
  Interventions: Biological: BOTOX

INTERVENTIONS:
Biological: BOTOX — 150 units of Botox injected intravaginally into the bulbocavernosum, pubococcygeus and puborectalis muscles along the lateral side walls, left and right as a one time injection under anesthesia.

SUMMARY:
The use of Botox injections intravaginally and progressive dilation under anesthesia has been shown to cure vaginismus. This study expands the use of Botox injections to include progressive dilation, post procedure supervised dilation and sex counseling to help women transition from dilators to intercourse. Since 2005 patients continue to experience a cure rate in excess of 90%. As of December 2012 more than 200 vaginismus patients have been treated this way.

In this completed study of 30 patients with a minimum of one year follow-up 29 vaginismus patients were able to advance to pain free intercourse (97%) and one patient failed to achieve her goals presumably due to uncontrolled anxiety relating to vaginal penetration.

DETAILED DESCRIPTION:
Vaginismus is the most common reason for unconsummated marriages. The more severe forms of vaginismus are often refractory to a variety of treatments such as Kegel exercises, dilator therapy, psychotherapy, sex counseling physical therapy, hypnotherapy, biofeedback, anti-depressants, anti-anxiety drugs, hymenectomy and vestibulectomy. In the larger cohort of 200 patients, a detailed data analysis of 150 patients (paper submitted) the average length of time of failed treatments was more than 7 years. 25% of vaginismus women suffered with this condition for more than a decade.

Spasm of the vaginal muscles is well defined in the scientific literature, first described by Sims in his 1861 report, as well as Lamont in 1978 and currently included in the DSM-IV definition of vaginismus. Pacik has reported on the prevalence of spasm of the bulbocavernosum, especially in the more severe forms of vaginismus, consistent with the history that intercourse feels like it is "hitting a wall", also noted by Lamont. The use of Botox injections as a treatment for vaginismus dates back to 1997. Since then several reports, including papers and presentations from our practice, have shown the efficacy of Botox injections for vaginismus. Botox is a very safe drug when used correctly. As of December 2012 more than 200 patients have been treated in our practice, mostly the more severe forms of vaginismus, who have been refractory to other forms of therapy. In this population dating back to 2005, the cure rate is in excess of 90%. There have been three minor complications of mild stress incontinence all of which resolved after about four months when the Botox was no longer active. One patient in this large cohort developed excessive vaginal dryness, likely due to block of the parasympathetic nerves which govern "letdown". Several patients have become pregnant and delivered normal children by vaginal childbirth.

The program to cure vaginismus is more than just injecting Botox under anesthesia and incorporates the following additional essential steps:

The areas of maximum spasm of the vaginal muscles are identified under sedation to determine where the Botox should be injected. The injections done under anesthesia are followed by additional injections of a long acting local anesthetic bupivacaine. After this the vagina is progressively dilated while the patient is still under anesthesia, and the dilators are further coated with a topical anesthetic. All these measures allow the patient to wake up in the recovery room with the large dilator in place and no discomfort. Following this, supervised dilation continues so that the patient becomes comfortable moving the dilator in and out of the vagina. This supervised dilation continues for a total of two to three mornings. During this time counseling is done with the couple to help instruct the correct use of the dilators, transition from dilators to intercourse, positions of pelvic floor relaxation and couple's counseling. Written instructions are given as well as a DVD addressing these aspects and close follow up and support by phone and email to ensure success of the program.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant healthy females aged 20-40 with Lamont level 1-4 primary vaginismus.
2. Willing to practice a reliable method of contraception for the first 4 months after treatment.
3. Able to understand and comply with the requirements of the study and sign Informed Consent.

Exclusion Criteria:

1. Female subjects who are pregnant (positive urine pregnancy test), trying to become pregnant, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
2. Allergy or sensitivity to any component of the test medication
3. History of poor cooperation, non-compliance with medical treatment, or unreliability.
4. Intact hymen, dyspareunia, secondary vaginismus, vulvodynia, dermatopathology of the vulva or perineum, anal fissure, associated urinary or rectal problems, complex pain disorders of the urogenital diaphragm or pelvic floor including pudendal nerve entrapment, psychiatric illness.
5. Treatment with botulinum toxin of any serotype prior to enrollment in study.
6. Any medical condition that may put the subject at increased risk with exposure to BOTOX including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function.
7. Evidence of alcohol, drug abuse or other relevant neuropsychiatric condition.
8. Infection or skin disorder at an anticipated injection site.
9. Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
10. Participation in an investigational drug study within 30 days of the Baseline Visit.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Pacik, MD, Principal Investigator — Plastic Surgery PA
Locations (1):
- Plastic Surgery Professional Association, Manchester, New Hampshire, United States

REFERENCES:
- [Background] Pacik PT. Botox treatment for vaginismus. Plast Reconstr Surg. 2009 Dec;124(6):455e-456e. doi: 10.1097/PRS.0b013e3181bf7f11. No abstract available. PMID 19952618
- [Background] Pacik PT. Vaginismus: review of current concepts and treatment using botox injections, bupivacaine injections, and progressive dilation with the patient under anesthesia. Aesthetic Plast Surg. 2011 Dec;35(6):1160-4. doi: 10.1007/s00266-011-9737-5. Epub 2011 May 10. PMID 21556985
- [Background] Pacik PT, Cole JB. When Sex Seems Impossible. Stories of Vaginismus & How You Can Achieve Intimacy. Odyne Publishing 2010
- [Background] Pacik PT. Understanding and treating vaginismus: a multimodal approach. Int Urogynecol J. 2014 Dec;25(12):1613-20. doi: 10.1007/s00192-014-2421-y. Epub 2014 Jun 4. PMID 24894201
- [Result] Pacik PT, Geletta S. Vaginismus Treatment: Clinical Trials Follow Up 241 Patients. Sex Med. 2017 Jun;5(2):e114-e123. doi: 10.1016/j.esxm.2017.02.002. Epub 2017 Mar 28. PMID 28363809
- [Result] Pacik, P. T. (2015), OnabotulinumtoxinA as Part of a Multimodal Program to Treat Vaginismus. Journal of Applied Biobehavioral Research, 20: 25-36. doi:10.1111/jabr.12037

RESULTS

PARTICIPANT FLOW:
Groups:
- BOTOX: Intravaginal (lateral aspects-bulbospongiosum) Botox injections, bupivacaine injections to the side walls of the vagina (cervix to introitus), progressive dilation under anesthesia and post procedure counseling and support to cure vaginismus.
  BOTOX: 150 units of Botox, and bupivacaine injected intravaginally into the bulbocavernosum, pubococcygeus and puborectalis muscles along the lateral side walls, left and right as a one time injection under anesthesia.
Period: Overall Study
Arm/Group | BOTOX
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BOTOX
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: years] | 27.3 [20 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Ability to Achieve Pain Free Intercourse.
Description: Patients need to be able to transition from the use of vaginal dilators to pain free intercourse, or to be able to continue using the #5 or #6 of 6 dilators in the absence of a partner.
Time Frame: one year
Measure: Number; unit: percentage of participants
Arm/Group | BOTOX
Number analyzed (Participants) | 31
percentage of participants | 90.3

ADVERSE EVENTS:
Arm/Group | BOTOX
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes